CLINICAL TRIAL: NCT06805435
Title: Is Continuous Non-Invasive Monitoring Accurate When Used on the Lower Extremity?: a Pilot Study
Brief Title: Is Continuous Non-Invasive Monitoring Accurate When Used on the Lower Extremity: Finger Vs Toe?
Status: Completed | Type: Observational
Sponsor: Riverside University Health System Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Baker, Research Coordinator, Riverside University Health System Medical Center
Other Study IDs: 2219626-3
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Validation; Blood Pressure; Device
Keywords: Acumen IQ cuff; continuous non-invasive blood pressure monitoring; Toe

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Healthy volunteers: Healthy volunteers consisting of medical students and residents at our institution.
  Interventions: Device: Continuous non-invasive blood pressure monitoring

INTERVENTIONS:
Device: Continuous non-invasive blood pressure monitoring — A continuous non-invasive blood pressure monitoring cuff will be placed on the volunteers index finger (as intended) and 2nd toe (primary outcome).

SUMMARY:
The goal of this observational study is to assess the validity of a continuous non-invasive blood pressure monitoring device, Acumen IQ cuff (Edwards Lifesciences LLC, Irvine, CA), when used on the toe in healthy volunteers. The main questions it aims to answer is:

• Can a continuous non-invasive blood pressure monitoring device accurately measure hemodynamic parameters when placed on a toe as compared to the finger in a healthy volunteer?

Secondary Outcomes:

* What are the effects of length and circumference of the middle phalanx of the 2nd toe on the accuracy of the Acumen IQ cuff (Edwards Lifesciences LLC, Irvine, CA) measurements compared to the measurements taken from the finger?
* What are the effects of a Valsalva maneuver on the measurements taken from the Acumen IQ cuff (Edwards Lifesciences LLC, Irvine, CA) on a toe compared to the Acumen IQ cuff (Edwards Lifesciences LLC, Irvine, CA) placed on the finger.

Participants will:

* Have blood pressures taken using an automatic blood pressure cuff (both arms and both calves)
* Have a continuous non-invasive blood pressure monitoring sensor placed on their finger and toe simultaneously for 10 minutes
* Be asked to valsalva briefly to induce a change in blood pressure to be observed by the dual sensors

DETAILED DESCRIPTION:
For each volunteer the investigators will measure the length from the proximal interphalangeal (PIP) joint to the distal interphalangeal (DIP) joint of the 2nd toe as well as the circumference at the center of the middle phalanx of the 2nd toe which the Acumen IQ cuff (Edwards Lifesciences LLC, Irvine, CA) will be placed on. Data including the hemodynamic measurements from the toe and finger cuffs will be collected. Laterality of cuff placement on finger and toes will be noted. Age, gender, height, and weight of the volunteers will be recorded.

During the trials the monitors will not be visible once necessary adjustments have been made and before data collection has begun. The two data sets from each sensor (finger and toe) will be linked together at the time of data collection. The investigators will not be able to tell which volunteer the data belongs to when analyzing the data.

Prior to the placing the Acumen IQ cuff (Edwards Lifesciences LLC, Irvine, CA), baseline blood pressures will be taken at the start of the study from each extremity using an automatic blood pressure cuff.

The healthy volunteer will have one Acumen IQ cuff (Edwards Lifesciences LLC, Irvine, CA) placed on the 2nd toe and one Acumen IQ cuff (Edwards Lifesciences LLC, Irvine, CA) place on the index finger. The study will be performed in a break room with minimal external stimulus. The volunteer will be asked to lie supine for approximately 3 minutes until the sensors have calibrated. They will remain in the supine position for another 5 minutes for data collection. An automatic blood pressure cuff on the contralateral lower extremity to the Acumen IQ cuff (Edwards Lifesciences LLC, Irvine, CA) will measure blood pressures at 0, 2.5, and 5 minutes. They will then be asked to perform a Valsalva maneuver at their own discretion for no longer than 5 seconds. The research protocol will be performed by the research coordinator on staff. Data collection occurs automatically every 20 seconds, but manual recording of data will be performed. The two continuous monitoring devices will be synced at the beginning of the study by simultaneously inputting a flagged event from which the start time will be inferred during data analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Medical student or resident

Exclusion Criteria:

* Medical history of Raynaud's or peripheral vascular disease
* Allergy to adhesive

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consistent of a convenience sample of available healthy volunteer medical students or residents.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Comparison between output from the continuous non-invasive blood pressure cuff placed on the volunteers index finger compared to the output from the continuous non-invasive blood pressure cuff placed on the volunteers 2nd toe. | Continuous non-invasive blood pressure measurements will be collected for 10 minutes
  The continuous non-invasive blood pressure cuff measures mean arterial pressure which will be compared between the index finger and 2nd toe of the same volunteer.

SECONDARY OUTCOMES:
Effects of length and circumference of the middle phalanx of the 2nd toe on the accuracy of the continuous non-invasive blood pressure cuff measurements compared to the measurements taken from the index finger. | Continuous non-invasive blood pressure measurements will be collected for 10 minutes.
  To compare the measurements from the index finger cuff to the 2nd toe cuff based on the length and circumference of the middle phalanx of the 2nd toe.
Validity of the continuous non-invasive blood pressure monitoring cuff on the toe compared to automatic blood pressure cuff measurements on the contralateral lower extremity. | Continuous non-invasive blood pressure measurements will be collected for 10 minutes
  To compare and assess the validity of the continuous non-invasive blood pressure monitoring cuff on the 2nd toe compared to measurements taken via an automatic blood pressure cuff from the contralateral lower extremity.

CONTACTS AND LOCATIONS:
Locations (1):
- Riverside University Health System Medical Center, Moreno Valley, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan is in place to share IPD at this time.